CLINICAL TRIAL: NCT06951867
Title: An Observational Multi-Country Post-Authorisation Safety Study to Evaluate the Risk of Serious Adverse Cardiovascular Events in Adolescent and Adult Patients With Severe Asthma Taking Tezepelumab
Brief Title: Tezspire Cardiac Events PASS
Acronym: TRESPASS
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: IQVIA Pvt. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00024
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Events; MACE
Keywords: post Marketing Requirements (PMR) study; cardiovascular events; non-fatal myocardial infarction; non-fatal stroke; cardiovascular death; arrythmias; coronary artery disease; heart failure; myocardial disorders
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure | interventions — tezepelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- tezepelumab severe asthma patients: patients with a diagnosis of severe asthma receiving tezepelumab
  Interventions: Drug: Tezepelumab
- tezepelumab unexposed asthma patients: patients with a diagnosis of severe asthma receiving non-tezepelumab standard of care for severe asthma

INTERVENTIONS:
Drug: Tezepelumab — The exposure of primary interest is tezepelumab for severe asthma. Exposure will be assessed based on prescriptions or administrations depending on the data source. A comparable cohort of unexposed patients treated with high-intensity SOC will be identified based on the presence of a trigger exposure (i.e., augmentation or change of the non-biologic high-intensity treatment that does not represent treatment de-escalation) to mirror tezepelumab start in the exposed cohort. Due to the limited knowledge of the cardiovascular profile of biologics, SOC for comparative analyses will only include non-biologic high-intensity treatment.
  Other Names: TEZSPIRE
  Groups: tezepelumab severe asthma patients

SUMMARY:
The aim of this study is to evaluate the risk of serious adverse cardiovascular events in adolescent and adult patients with severe asthma taking tezepelumab compared to a population receiving standard of care treatment for severe asthma.

DETAILED DESCRIPTION:
Tezepelumab (brand name: TEZSPIRE®), a human monoclonal antibody specific for the epithelial cell-derived cytokine thymic stromal lymphopoietin (TSLP), was recently launched as a first-in-class biologic add on treatment for patients with severe asthma. Results from DESTINATION, a long-term extension, phase 3 trial, showed a numeric imbalance in the occurrence of cardiac disorder system organ class serious adverse events (SAEs) in participants receiving tezepelumab compared to placebo. The observed imbalance resulted in the inclusion of serious cardiovascular events as an important potential risk to be addressed in the European Union (EU) risk management plan (RMP). AstraZeneca proposed to evaluate the risk of serious cardiovascular events with long-term tezepelumab treatment to meet regulatory requirements under a category 3 Post-Authorisation Safety Study (PASS).

This study is a non-interventional, longitudinal, population-based cohort study, using secondary data derived from multiple data sources. The study will consist of descriptive and a prevalent new-user design for comparative analyses of serious cardiovascular events outcomes in adolescent and adult patients with severe asthma exposed and unexposed to tezepelumab.

The study will be conducted using data sources from Denmark, France, Germany, and the United States of America (USA). The start of the study period will correspond to tezepelumab market launch date in each country of interest (i.e. between Q1 2022 - Q3 2023). An approximately five-year study period is planned in each country, with an anticipated last date of study period on 28 February 2029.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of asthma receiving tezepelumab or high-intensity SOC treatment for severe asthma at any point during the study inclusion period.

Exclusion Criteria for both exposed and unexposed groups include:

* <12 months of data availability prior to index date,
* age <12 years at index date,
* history of congenital heart disease or heart transplant outcome-specific exclusion criterion applied for each objective will include the presence of non-fatal myocardial infarction or stroke and the specific outcome of interest in the 180 days prior to index date
* for comparative analysis, an additional exclusion criterion will be considered, i.e. exposure to non-tezepelumab biologics on index date or within the 5-half-life clearance period of the biologic
* matching criteria (including, among other variables, the type and duration of SOC exposure in the 12 months before index date and propensity score [PS] matching) will be applied to ensure exposed and unexposed patients' comparability

Ages: 12 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted using data sources from Denmark, France, Germany, and the United States of America (USA).
  The source population will consist of patients with a diagnosis of asthma receiving tezepelumab or high-intensity SOC treatment for severe asthma at any point during the study inclusion period. From this source population, the exposed study population (i.e. patients who initiate tezepelumab treatment) and the unexposed study population (i.e. comparable patients who are unexposed to tezepelumab) will be identified.
Sampling Method: Probability Sample
Enrollment: 95574 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
composite outcome MACE | five years from tezepelumab market launch
  The primary outcome of interest is the composite outcome MACE, consisting of non-fatal myocardial infarction, non-fatal stroke, or cardiovascular death.

SECONDARY OUTCOMES:
composite of four serious adverse cardiovascular events | five years from tezepelumab market launch
  The secondary outcomes of interest are a composite of four serious adverse cardiovascular events, including arrhythmias, coronary artery disease, heart failure and myocardial disorders, and the individual components of the primary and secondary composite outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Egger, Principal Investigator — Iqvia Pty Ltd
Locations (4):
- Healthcare Integrated Research Database (HIRD), Wilmington, Delaware, United States
- Danish registries (access/analysis), Copenhagen, Denmark
- French National Health Data System (SNDS), Paris, France
- Team Gesundheit GKV Claims data (SHI), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved, AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/